CLINICAL TRIAL: NCT04171804
Title: Efficacy of Prefrontal Transcranial Direct Current Stimulation On Cognitive Functions and Electrophysiological Measures In Parkinson's Disease Mild Cognitive Impairment
Brief Title: Efficacy of Transcranial Direct Current Stimulation In Parkinson's Disease MCI
Acronym: PDMCIStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Serkan Aksu, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-055
Record Dates: First submitted 2019-11-03; First posted 2019-11-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Mild Cognitive Impairment; Transcranial Direct Current Stimulation; Cognitive functions; Electrophysiology; Event related potentials
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Left anodal/right anodal transcranial direct current stimulation over the dorsolateral prefrontal cortex
  Interventions: Device: Transcranial direct current stimulation
- Sham (Sham Comparator): Sham transcranial direct current stimulation over the dorsolateral prefrontal cortex
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Participants will receive a total of 10 stimulation sessions on 5 consecutive days (twice a day with 3-4 hours interval). During each session, 2 milliAmpers (mA) of active or sham tDCS will be applied for 20 minutes over the dorsolateral prefrontal cortex (left anodal/right anodal).
  Other Names: tDCS; Direct current stimulation; transcranial electrical stimulation

SUMMARY:
The aim of the present study is to investigate the efficacy of prefrontal transcranial Direct Current Stimulation (tDCS) on cognitive functions and electrophysiological measures in Parkinson's Disease Mild Cognitive Impairment (PD-MCI). The participants will be assigned to active and sham groups (1:1) and will receive 10 sessions of tDCS (twice a day) for 5 days. The study will also examine if the effects may last for a month. The participants will be assigned to active and sham groups (1:1) and will receive 10 sessions of tDCS (twice a day) for 5 days. The study will also examine if the effects may last for a month.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is the second most common neurodegenerative disorder. The period that apparent cognitive deficits exist without disrupting daily life activities is named as Mild Cognitive Impairment (PD-MCI). Treatments were considered to be more efficacious in PD-MCI than PD dementia as relatively less permanent changes in cortical structures occured. No approved treatments exist in PD-MCI and non-pharmacological treatments are under investigation as drugs have considerable amount of adverse effects.

Event Related Potentials (ERP) measurements have the advantages of providing direct and objective evidence of central nervous system functions, imaging of the activity of the cortical areas and being unaffected by motor deficits. ERP parameters were found to be related to cognitive functions and disrupted in PD and PD-MCI. Thus, ERP parameters were suggested to be useful in treatment efficacy assessment.

Transcranial Direct Current Stimulation (tDCS) is a promising non-invasive brain stimulation method. Ameliorating effects of tDCS on cognition and ERPs were observed. Enhancing effects of tDCS on some cognitive deficits were also reported in PD.

Few studies reported the efficacy of both tDCS and physical therapy/cognitive training and none assessed the efficacy of tDCS solely, compared to a sham control group. All studies assessed the efficacy without using electrophysiological measurements that reflect central nervous system functions directly. In this project, the efficacy of tDCS will be compared to a sham tDCS group and be assessed with electrophysiological measurements for the first time.

The study is a double-blind randomized controlled trial. The sample will be consisted of twenty six participants diagnosed as having PD-MCI due to Movement Disorders Society Level 2 criteria. The participants will be assigned to active or sham groups. Then, neuropsychological test performances and ERP parameters during Oddball paradigm and Continuous Performance Test will be measured. Then, participants will be applied ten active or sham sessions of left anodal/right cathodal tDCS over the dorsolateral prefrontal cortex (DLPFC). All measurements will be repeated both immediately and 1-month after the applications.

Succinctly, the aim of this project is to assess the effect of ten sessions left anodal/right cathodal tDCS over the DLPFC on cognitive functions and electrophysiological parameters in PD-MCI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD with at least two of the four diagnostic criteria for PD (tremor, rigidity, bradykinesia, and postural instability) in accordance with the United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria, issued by a neurologist specializing in movement disorders;
* Disease staging between I and III, according to the modified Hoehn and Yahr scale;
* Clinical diagnosis of PD- MCI in accordance with Level 2 Movement Disorders Society- Task Force diagnostic criteria;
* An unchanged stable and optimal regimen of dopaminergic medication for at least one month before study entry and able to continue on a stable regimen for the duration of the study;
* Ability to provide written informed consent;
* 5 or more years of education;
* Right-hand dominancy;
* Not taking any psychoactive medications before the previous month of the study and for the duration of the study;
* Naïve to tDCS.

Exclusion Criteria:

* Diagnosis or evidence of secondary or atypical parkinsonism;
* Patients with dementia;
* Less than 5 years of education;
* Previous history of surgical intervention for PD such as deep brain stimulation (DBS);
* Diagnosis of active major depressive disorder, psychotic disorders, bipolar disorder, alcohol use disorder and substance use disorders;
* Any history of any clinically significant neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, multiple sclerosis, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes;
* Significant hearing loss or visual impairment;
* Diagnosis of any serious or uncontrolled medical condition such as chronic obstructive pulmonary disease, congestive heart failure or renal failure;
* Skin diseases that could potentially cause irritations under electrodes
* Patients missing two consecutive protocol sessions;
* Illiteracy, deficient language or refusal to participate or being not able to follow instructions or complete study tasks;.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Changes in response conflict in the Stroop Test during the study period | Up to one month
  The stroop effect consists of the semantic and the response conflict. Response conflict (time in milliseconds) is obtained by subtracting the semantic conflict (time in milliseconds obtained in the second step of the protocol) from the stroop effect (time in milliseconds obtained in the first step of the protocol). Minimum time difference is 0 and maximum time difference is 100 milliseconds. Lower time differences indicate better performance and higher time differences indicate worse performance.
Change in the verbal fluency performance during the study period | Up to one month
  Verbal fluency is a test that measure multiple domains of cognition such as executive functions and language functions. Letter Verbal Fluency assesses the number of words beginning with certain letters that participants can generate within 60 seconds, the Category Verbal Fluency assesses the number of words within particular categories participants can generate within 60 seconds. Minimum score is 0 and maximum score is 80. Lower scores indicate worse performance and higher scores indicate better performance.
Changes in Trail Making A Test performance during the study period | Up to one month
  Trail Making A Test is a widely used as a quick and easy to administer measure of attention. Lower reaction times indicate better performance and higher reaction times indicate worse performance. Minimum time is 10 milliseconds and maximum time is 150 milliseconds.
Changes in digit span during the study period | Up to one month
  The Digit Span test is a measure of verbal short-term/working memory. Subjects must recall all digits either in forward (digit span forward) or backward (digit span backward) order.
  Digit span forward total score: 0-10; higher score indicate better performance, digit span backwards total score: 0-10; higher score indicate better performance
Changes in delayed recall performance during the study period | Up to one month
  Memory performance was assessed using delayed recall (number of units recalled) on the Wechsler Memory Scale (WMS-IV) logical memory (story recall) test. Scores represent a sum of recalled units of two different stories after a 30 minute delay. Total scores range from 0 to 50 (0-25 for each story) with higher scores reflecting better memory performance.
Changes in verbal memory processes performance during the study period | Up to one month
  The Verbal Memory Processes Test is a 15-word word-list learning test with a 40-minute delayed recall addition based on the Rey Auditory Verbal Learning Test which gives the opportunity to evaluate the processes of working memory, learning or acquiring knowledge, retention of information, and recalling.
  It consists of immediate recall, learning score and a 40-min delayed recall test, followed by total recall. Higher scores indicate better performance in all indexes of the test. Minimum scores are 0 and maximum scores are 15 for immediate recall, delayed recall and total recall and 150 for learning score, respectively.
Changes in face recognition performance during the study period | Up to one month
  Benton Facial Recognition Test is a common test assessing visuo-spatial functions. It was developed by Benton in 1969. It is standardized to determine the capacity to identify and distinguish unrecognized human faces. This test consists of 22 pages of A4 size and there are face pictures on these pages. Only one page of pages is numbered. There is a stimulant picture on pages with no page numbers. Numbered pages have 6 pictures to select from among the responses. The application period of the test is 5-15 minutes and the time factor is not evaluated separately. Higher scores indicate better performance and lower scores indicate worse performance. Minimum score is 0 and maximum score is 54.
Changes in judgment of line orientation performance during the study period | Up to one month
  A test of visuospatial judgement. The test measured the participant's ability to match the angle and orientation of lines in space. There were 30 trial in total. Correct response in a trial was awarded one point. Minimum score is 0 and maximum score is 30. Higher scores represent better performances.
Changes in the naming performance during the study period | Up to one month
  The naming performance will be measured by the Boston Naming Test Short Form and Responsive Naming Test. Boston Naming Test consists of 45 pictures to be named. Minimum score is 0 and maximum score is 45. Higher scores indicate better performance and lower scores indicate worse performance. In the Responsive Naming Test, participants answer the questions such as "What do women apply to their lips?" Minimum score is 0 and maximum score is 10. Higher scores indicate better performance and lower scores indicate worse performance.
Changes in amplitudes (in microvolts) for parameters from the ERP tests during the study period for parameters from the ERP tests during the study period | Up to one month
  Amplitudes (in microvolts) for the following parameters from the ERP tests will be collected as primary endpoints:N1, P3 and other common wave forms for both Two-tone auditory oddball paradigm and Continuous Performance Test ERP paradigms.
Changes in detection sensitivity from the behavioral responses during the Two-tone auditory oddball and Continuous Performance Test ERP paradigms during the study period | Up to one month
  Detection sensitivity from Signal Detection Theory (d', calculated as [zFA - zHR], where z is the inverse of the standard normal cumulative distribution, FA is the false-alarm rate [the proportion of responses made to stimuli that were not targets], and HR is the hit rate [the proportion of correct identifications of target stimuli]) during the Two-tone auditory oddball and Continuous Performance Test ERP paradigms will be measured.
Changes in reaction times from the behavioral responses during the Two-tone auditory oddball and Continuous Performance Test ERP paradigms during the study period | Up to one month
  Reaction times for the correct behavioral responses during the Two-tone auditory oddball and Continuous Performance Test ERP paradigms will be measured.

SECONDARY OUTCOMES:
Correlation between changes in behavioral measures and changes in amplitudes of ERP components | Up to one month
  Correlation between changes in detection sensitivity from the behavioral responses and changes in amplitudes of ERP components during the Two-tone auditory oddball and Continuous Performance Test ERP paradigms during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Aksu, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No